CLINICAL TRIAL: NCT00259103
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Safety, Pharmacokinetics and Efficacy of Intravenous Recombinant Human Relaxin (rhRlx) in Pregnant Women Scheduled for Induction of Labour
Brief Title: Recombinant Human Relaxin (rhRlx) in Pregnant Women Scheduled for Induction of Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corthera, Inc.(formerly BAS Medical, Inc.), a member of the Novartis group of companies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLX.CR.001
Record Dates: First submitted 2005-11-15; First posted 2005-11-29 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Labor, Induced
Keywords: relaxin; pregnancy; cervical ripening; normal pregnancy at least at 40 weeks of gestation
MeSH Terms: interventions — serelaxin protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 7.5 µg/kg/d (Experimental): Participants who received intravenous (IV) infusion of 7.5 µg/kg/d serelaxin, all during part A.
  Interventions: Drug: Serelaxin
- 25 µg/kg/d (Experimental): Participants who received intravenous (IV) infusion of 25 µg/kg/d serelaxin, all during part A.
  Interventions: Drug: Serelaxin
- 75 µg/kg/d (Experimental): Participants who received IV infusion of 75 µg/kg/d serelaxin, some during part A and others during part B.
  Interventions: Drug: Serelaxin
- Placebo (Experimental): Participants who received IV infusion of placebo, some during part A and others during part B.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Serelaxin
  Arms: 25 µg/kg/d; 7.5 µg/kg/d; 75 µg/kg/d
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of rhRlx for cervical ripening, when compared to a placebo.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled, dose escalation study of healthy female subjects at ≥ 40 weeks gestation and who are scheduled for induction. A dose-escalation portion of the study is followed by a randomized, double-blind, placebo-controlled portion of the study. The endpoints include cervical ripening, as well as progression to labor and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Normal pregnancy
* At least 40 weeks of gestation
* Otherwise healthy

Exclusion Criteria:

* Anemia or hypertension
* Presence of chronic disease
* Endometriosis
* Known fetal anomaly
* Substance abuse
* History of cancer

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2005-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Cervical ripening | Through 24 hours

SECONDARY OUTCOMES:
Progression to active labor and delivery | Within 7 Days of Drug Infusion

CONTACTS AND LOCATIONS:
Overall Officials: Sam Teichman, MD, Study Director — Chief Medical Officer of BAS Medical, Inc.
Locations (3):
- Russia (3):
  - Novosibirsk State Medical Academy, Novosibirsk
  - Evidence CPR, Saint Petersburg
  - D.O. Ott Research Institute of Obstetrics and Gynecology, Saint Petersburg

REFERENCES:
- [Derived] Weiss G, Teichman S, Stewart D, Nader D, Wood S, Breining P, Unemori E. Recombinant human relaxin versus placebo for cervical ripening: a double-blind randomised trial in pregnant women scheduled for induction of labour. BMC Pregnancy Childbirth. 2016 Sep 5;16(1):260. doi: 10.1186/s12884-016-1046-1. PMID 27596360